CLINICAL TRIAL: NCT02684773
Title: Impact Of In-Centre Nocturnal Hemodialysis On Cardiac Remodeling In End-Stage Renal Disease: A Long-Term Follow-Up Study
Brief Title: In-Centre Nocturnal Hemodialysis (INHD): A Long-Term Follow-Up Study
Acronym: INHD
Status: Completed | Type: Observational
Sponsor: Unity Health Toronto (Other)
Collaborators: Heart and Stroke Foundation of Canada (Other)
Responsible Party: Sponsor
Other Study IDs: G-14-0005856
Record Dates: First submitted 2016-01-07; First posted 2016-02-18 (Estimated); Last update posted 2017-04-26 (Actual); Status verified 2017-04

CONDITIONS: End-stage Renal Disease; Left Ventricular Hypertrophy
Keywords: Hemodialysis; Left Ventricular Mass; Cardiac Magnetic resonance Imaging
MeSH Terms: conditions — Kidney Failure, Chronic; Hypertrophy, Left Ventricular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum and Plasma sample collection
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Incentre Nocturnal Hemodialysis: These are patients who converted to incentre nocturnal hemodialysis (8 hours/session, 3 sessions/week) from conventional hemodialysis (4 hours/session, 3 sessions/week) at the inception of this study and are eligible for the long-term follow-up phase of the study.
  Interventions: Procedure: In-centre Nocturnal Hemodialysis
- Conventional Hemodialysis: These are patients treated with conventional hemodialysis (4 hours/session, 3 session/week) who elected to remain on this dialysis schedule at the inception of this study and are eligible for the long term follow-up phase of the study.
  Interventions: Procedure: Conventional Hemodialysis

INTERVENTIONS:
Procedure: Conventional Hemodialysis — The intervention involves 3 hemodialysis sessions/week that consists of 4 hours/session
  Groups: Conventional Hemodialysis
Procedure: In-centre Nocturnal Hemodialysis — The intervention involves 3 hemodialysis sessions/week administered overnight (8 hours/session) in-hospital
  Groups: Incentre Nocturnal Hemodialysis

SUMMARY:
Background: In 2010, approximately 39000 Canadians had end-stage renal disease (ESRD), and the prevalence rate of dialysis has increased by 189% over the past 2 decades. The annual mortality rate remains high at ~15%, and cardiovascular events are the leading cause of death. Intensification of conventional dialysis schedules has been the major focus in recent years. Currently, most Canadian dialysis patients receive conventional in-center hemodialysis (CHD), which is administered as a 3-4 hour session 3/week. Recent research has focused on home nocturnal hemodialysis (8 hours of hemodialysis at home for 5-6 nights/week), which may have substantial cardiovascular benefits, including regression of left ventricular (LV) hypertrophy, improved LV ejection fraction and enhanced blood pressure control. Nevertheless, this dialysis modality is only feasible in a highly selected minority of ESRD patients who can self-manage their dialysis treatment at home. In-center nocturnal hemodialysis (INHD), administered as 7-8 hours of hemodialysis in hospital for 3nights/week, represents a promising and practical alternative for many dialysis patients. In a Canadian Institutes for Health Research (CIHR) supported cohort study, the investigators have recruited 67 patients and have completed 1-year follow-up. There is a compelling need for longer-term follow-up, since all the published randomized controlled trials are of short duration (6-12 months), while renal replacement therapy is a life-long treatment. Furthermore, the observed large variability of cardiac remodeling in individual ESRD patients remains poorly understood. Therefore, the current study is an extended follow-up phase (5 years from enrollment) on the completed 1-year follow-up period and the purpose of this study is to objectively evaluate the long-term effects of more intensified hemodialysis treatment which the INHD modality offers.

Need for Long-term and Generalizable Data: In contrast to the seminal Alberta trial which showed a significant LV mass reduction with home nocturnal hemodialysis, the recently reported Frequent Hemodialysis Network Nocturnal Trial demonstrated only a trend toward reduction in LV mass. It is likely that the highly selected participants, inadequate trial power and duration (12 months) account for the observed results. Currently, it is unknown whether INHD, which is less intensive but more feasible for most ESRD patients, is associated with similar cardiovascular benefits in the long term.

Objective:

1. To determine the long-term effects of INHD on (i) LV mass; (ii) global and regional LV systolic and diastolic function; (iii) myocardial tissue characteristics; (iv) left atrial structure and function; (v) selected cardiovascular biomarkers in ESRD patients.
2. To examine the determinants and mechanisms of cardiac remodeling in ESRD

Hypothesis: Conversion to INHD is associated with sustained improvements in cardiovascular structure and function, as compared to conventional hemodialysis (CHD) in patients with end-stage renal disease (ESRD).

Study Design and Population: This will be a 2-centre, prospective, longitudinal cohort study of 67 adult ESRD patients (INHD subjects and CHD controls) enrolled in the original study. All eligible participants who provide consent will undergo cardiac Magnetic Resonance Imaging (MRI) examination and bloodwork at 5 years since enrollment in the study. Other follow-up procedures include the following -electrocardiogram, transthoracic echocardiogram, ambulatory blood pressure monitoring, lateral x-ray of the aorta, and completion of questionnaires.

Outcome: The primary endpoint is the change in LV mass over 5 years, as measured by cardiac MRI. Secondary endpoints include LV size, global and regional diastolic and systolic function, left atrial size and function, changes in myocardial tissue characteristics, blood pressure, serum troponin, norepinephrine, Brain Natriuretic Peptide (BNP), high sensitivity C-Reactive Protein (hsCRP), interleukin-6, matrix metalloproteinases, fibroblast growth factor-23, fetuin-A, transforming growth factor-beta, connective tissue growth factor, clinical events, and quality of life.

Significance: The provision of an enhanced dialysis regimen has emerged as the most promising avenue through which to modify the dismal cardiovascular outcomes in patients receiving chronic hemodialysis. INHD represents a means of administering such therapy to a broad spectrum of dialysis patients for whom home therapies would not be feasible. This study will be the first to precisely define the long-term cardiac effects of intensified dialysis and to elucidate the mechanisms of cardiac remodeling in ESRD, using cardiac MRI and other novel biomarkers. These important observational findings may have a major impact on the optimal management and outcome of ESRD patients in the real world.

ELIGIBILITY:
Inclusion Criteria:

* all patients who were enrolled in the original one-year follow-up phase of the study and are eligible for the long-term follow-up phase

Exclusion Criteria:

* inability to provide informed consent for long-term follow-up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients who converted to in-centre nocturnal hemodialysis and their matched controls will be drawn from a population of prevalent chronic hemodialysis patients.
Sampling Method: Non-Probability Sample
Enrollment: 67 (Actual)
Dates: Start 2014-07; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Change in left ventricular mass index by cardiac MRI assessment | 5 years from Baseline procedure

SECONDARY OUTCOMES:
Changes in left ventricular end diastolic and systolic volume by cardiac MRI assessment | 5 years from baseline procedure
Changes in regional left ventricular systolic and diastolic function by cardiac MRI assessment | 5 years from baseline procedure
Changes in myocardial tissue characteristics by cardiac MRI assessment | 5 years from baseline procedure
Changes in blood pressure | 5 years from baseline procedure
Changes in quality of life | 5 years from baseline procedure
Changes in hs-CRP levels (mg/L) | 5 years from baseline procedure
Changes in BNP levels (ng/L) | 5 years from baseline procedure
Changes in serum troponin I levels (ug/L) | 5 years from baseline procedure

CONTACTS AND LOCATIONS:
Overall Officials: Ron Wald, MD, Principal Investigator — Unity Health Toronto; Andrew T Yan, MD, Principal Investigator — Unity Health Toronto
Locations (2):
- Canada (2):
  - St. Paul's Hospital, Vancouver, British Columbia
  - St. Michael's Hospital, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No